CLINICAL TRIAL: NCT01552148
Title: Randomized, Controlled, Observer-blinded Study on the Efficacy of TAP Block With 0.375% Levobupivacaine in Terms of PCA Morphine Postoperative Consumption in Patients Undergoing Laparoscopic Hysterectomy
Brief Title: Transversus Abdominis Plane Block for Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituti Ospitalieri di Cremona (Other)
Responsible Party: Principal Investigator, Giorgio Danelli, Chief of the Anaesthesia Department, Istituti Ospitalieri, Cremona, Istituti Ospitalieri di Cremona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5504/2012LD
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Hysterectomy; Laparoscopic Surgery

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Group TAP (US guided) (Active Comparator): 23 patients receiving bilateral US guided transversus abdominis plane block with 20ml of 0.375% levobupivacaine on each side, under general anaesthesia (TIVA), after induction and before surgical start
  Interventions: Other: USguided bilateral TAP block; Drug: Morphine Patient Controlled Analgesia
- Group Control (Other)
  Interventions: Drug: Morphine Patient Controlled Analgesia

INTERVENTIONS:
Other: USguided bilateral TAP block — 23 patients receiving bilateral US guided transversus abdominis plane block with 20ml of 0.375% levobupivacaine on each side, under general anaesthesia (TIVA), after induction and before surgical start
  Arms: Group TAP (US guided)
Drug: Morphine Patient Controlled Analgesia — Morphine PCA i.v. (bolus 2mg, lockout 8 min)
  Arms: Group TAP (US guided)
Drug: Morphine Patient Controlled Analgesia — Morphine PCA i.v. (bolus 2mg, lockout 8min)
  Arms: Group Control

SUMMARY:
Purpose To evaluate whether adding a transversus abdominis plane block in patients undergoing elective laparoscopic hysterectomy reduces Patient-controlled analgesia (PCA) morphine requirements during the first 24 hours postoperatively.

Forty-six patients undergoing laparoscopic hysterectomy will be randomized into two groups:

1. Group treatment TAP (n=23) will receive the following analgesia:

   * US guided transversus abdominis plane block performed with 40ml of 0.375% levobupivacaine (20 ml per side) after general anaesthesia induction, before surgical start
   * Morphine PCA with loading dose i.v. titrated by the PACU nurse if pain > 5/10 at rest
2. Group control will receive:

   * Morphine PCA with loading dose i.v. titrated by the PACU nurse if pain > 5/10 at rest

Primary Outcome Measures:

Morphine consumption (mg) (Time Frame: 24 hours) in Groups TAP and Control

Secondary Outcome Measures:

* Pain at rest and during movement quantified as Numerical Rating Scores (0-10) for pain when resting in bed and during cough during the first 24 hours postoperatively
* Time to PACU dimission, evaluated as patient's achievement of a White's score > or = 12/14
* Time to home discharge, evaluated as patient's achievement of a PADDS score > or = 9
* Functional patient capacity as measured before surgery and whenever a White's score > or = 12 will be reached (2minute walking test)
* Eventual side effects such as nausea/vomiting

DETAILED DESCRIPTION:
After the start of the study, we had a higher drop out size than expected. We therefore added a 13% of patient to initial power calculation to compensate for drop outs.

Total number of patients enrolled = 52 (46 + 6) Total number of patients who completed the study = 44

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age < 70 years
* ASA I - II - III
* undergoing elective laparoscopic hysterectomy
* signed informed consent

Exclusion Criteria:

* chronic therapy with opioids/ antidepressants
* surgical conversion to open abdominal hysterectomy
* urgent/emergent surgery
* postoperative transfer to the intensive care unit
* pregnancy or breast feeding
* known allergy to any drug medication
* local skin infection
* epilepsy
* high bilirubin level (> 3mg/dl) or high hepatic enzymes levels (> 250UI)
* high creatinin level (> 1.4mg/dl)
* 18Kg/m2 < BMI < 30Kg/m2
* alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
PCA morphine consumption in the two groups within the first 24 postoperative hours | 24 hours postoperatively

SECONDARY OUTCOMES:
Numerical Rating Scores for pain at rest and during movement | 24 hours postoperatively
Time to discharge from Recovery Room | 24 hours postoperatively
  Time to achieve a White's score > or = 12
time to discharge from the surgical floor | 24 hours postoperatively
  time to achieve a PADDS score > or = 9
evaluation of patients' functional capacity postoperatively versus baseline | 24 hours postoperatively
  2-minute walking test assessed as soon as a White's score > or = 12 has been reached or every 30minutes until patient is capable to walk
postoperative nausea/vomiting incidence | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona, CR, Italy